CLINICAL TRIAL: NCT06498557
Title: Results of Postoperative Analgesis Protocols Applied in Total Knee Arthroplasty:Observational Study
Brief Title: Postoperative Analgesis in Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Senay Canikli (Other)
Responsible Party: Sponsor-Investigator, Senay Canikli, MD, Samsun University
Organization: Samsun University (Other)
Other Study IDs: GOKAEK 2024/10/1
Record Dates: First submitted 2024-06-29; First posted 2024-07-12 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-07

CONDITIONS: Knee Arthroplasty
Keywords: POSTOPERATIVE PAIN; Knee Arthroplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group S: SFIP block will be applied for postoperative analgesic purposes
  Interventions: Other: Peripheral nerve block methods
- Group IP: SFIP block will be applied for postoperative analgesic purposes
  Interventions: Other: Peripheral nerve block methods

INTERVENTIONS:
Other: Peripheral nerve block methods — We apply different nerve blocks to patients for analgesic purposes after knee replacement surgery. These blocks are a combination of SFIP block and adductor channel block and iPACK block.

SUMMARY:
Postoperative analgesic treatment methods are applied to patients who have undergone knee arthroplasty. These applications are a routine part of the procedure. It is medically and ethically necessary. Postoperative analgesia applications are started during the intraoperative period and continued during the postoperative period. The analgesia protocol to be used is shaped by the characteristics of the patient and the skill and experience of the anesthesiologist. The scientifically accepted method is multimodel analgesia protocols. These protocols cover a wide range from paracetamol to opioids to peripheral and central blocks (methods such as suprainguinal fascia iliac block (SFIP), adductor block (ACB) and infiltration analgesia (IPACK) applied between the posterior elements of the knee and the popliteal artery). Our aim in this study is to evaluate the effects of analgesia protocols applied to patients undergoing knee arthroplasty surgery on inflammatory biomarkers (such as neutrophil lymphocyte ratio (NLR), platelet lymphocyte ratio (PLR), systemic immune inflammation score (SII), lactate) obtained from routine blood and blood gas examinations in the first 24 hours of the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* ASA I,II,III patients
* Patients who will undergo elective surgery

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients with bleeding diathesis
* Those who are allergic or sensitive to local anesthetics and opioid drugs,
* Those who use gabapentinoids
* Patients with neurocognitive disorders,
* Patients with chronic organ failure,
* Mothers with suspected pregnancy, pregnant or breastfeeding mothers
* Patients using opioids
* Those who use steroids
* Those with a history of substance use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among patients who had elective knee replacement surgery, those who underwent postoperative nerve block
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | postoperative 24 hours
  Pain levels of patients will be evaluated with the Numerical Pain Scale (NRS) in the first 24 hours postoperatively.

SECONDARY OUTCOMES:
inflammatory mediators | preoperative 24 hours
  NLR
inflammatory mediators | preoperative 24 hours
  PLR
inflammatory mediators | preoperative 24 hours
  SII
inflammatory mediators | preoperative 24 hours
  Lactate

CONTACTS AND LOCATIONS:
Overall Officials: Senay canikli adıgüzel, Study Director — Samsun University
Locations (1):
- SAMSUN UNIVERSITY Samsun Training and research hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants' data will not be shared. After the study is written as an article, it can be shared if the editor of the journal wishes